CLINICAL TRIAL: NCT06750367
Title: Effects of Klapp Method Exercises on Pain, Posture Correction and Self-efficacy in Breast Feeding Females With Kyphotic Posture
Brief Title: Effects of Klapp Method Exercises in Breast Feeding Females With Kyphotic Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0526
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Postural; Defect; Breast Feeding
Keywords: exercises; pain; posture; female; self-efficacy
MeSH Terms: conditions — Breast Feeding; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Klapp method exercises (Experimental): Four pointwalk followedby twopointwalk&backwalk: This exercise is basic, it is a mobility exercise and always applied at the beginning of the program. Breathing exercise from a kneeling position: (raising hands with inhalation lowering hands with exhalation). Simple bounce glide with simultaneous breathing: (a stretching,strengthening and corrective exercises) Bunny hop: (for stretching and strengthening). Greeting: (Stretching and mobilization of thalamus)
  Interventions: Other: Klapp method exercises
- At-Home exercises program (Active Comparator): The researcher will prescribe stretching of neck, upper limb and thoracic region of participants as a baseline treatment. The control group will continue with their normal activities and pain relief methods. Additionally, they will be given printed information on an at-home exercise program, such corrective exercises (Chin tuck, stretching of neck extensor muscles and pectoral muscle groups in standing and supine positions) (16), posture correction exercises (This exercise program consisted of 2 strengthening (of the deep cervical flexors and shoulder retractors), and breathing exercises (Deep breathing is an exercise that can regulate breathing patterns and improve posture. The deep breathing that is done repeatedly can overcome stiffness in the thoracic cage and straighten the curve of thoracic kyphosis).They will be asked to perform the period of 1-month twice in a week for 50 min with10 repetitions of each exercise
  Interventions: Other: At-Home exercise program

INTERVENTIONS:
Other: Klapp method exercises — The researcher will administer Klapp method exercises to the participant for a period of 1 month (twice in a week for 50 min .The researcher will perform stretching of upper limb, neck and thoracic region to the participants as a baseline treatment. Klapps exercises program include four point walk followed by two point walk and back walk, breathing exercise from kneeling position, breathing exercise from quadrapedal position, simple bounce glide with simulanteos breathing, bunny hop greeting. Each exercise will be performed with 10 repetitions
  Arms: Klapp method exercises
Other: At-Home exercise program — theywill begiven printed information on an at-home exercise program, such corrective exercises (Chin tuck, stretchingof neck extensormuscles andpectoral musclegroups instandingandsupinepositions) (16) ,posturecorrection exercises(Thisexerciseprogramconsistedof2strengthening(of thedeep cervical flexorsandshoulderretractors)(26) ,andbreathingexercises(Deep breathing is an exercise that can regulate breathing patterns and improve posture. The deep breathing that is done repeatedly can overcome stiffness in the thoracic cage and straighten the curve of thoracic kyphosis)(27).Theywillbeaskedtoperformtheperiodof1month twiceinaweekfor50minwith10repetitionsofeachexercise.
  Arms: At-Home exercises program

SUMMARY:
Group A will be given Klapp method exercises to the participant for a period of 1 month twice in a week for 50min. Group B will be given printed information on an at-home exercise program, such, posture correction,corrective exercises and breathing exercises. They will be asked to perform the exercises twice weekly during the study and follow-up period. All these sessions will be of 50 minute for 2 session per week for 4 weeks

DETAILED DESCRIPTION:
The Klapp exercises program, is an active therapeutic exercise that aims to stretch, mobilize, and strengthen the spine, offering both pain reduction and postural improvement. This method is widely applied, for the correction of vertebral deformities such as kyphosis, lordosis and scoliosis, to the treatment of thoracic cage abnormalities and thoracic cage shape changes after thoracoplasty, as well as in the treatment of spinal muscle interference from polio and spinal osteochondrosis.

The aim of this study to investigate the effects of klapp method exercises on pain, posture correction and self-efficacy in breast feeding females with kyphotic posture.

This will be a randomized Controlled trial conducted on (32) participants. Data will be collected from Civil hospital and Al-siddique hospital, Sialkot by using non-probability convenience sampling technique. Breast feeding females between the age of 22 to 30 with kyphotic posture. Participants who had a history orthopedic disorder, orthopedic surgery, history of recent fracture, non-lactating females will be excluded from this study. A sample of (32) will be divided in to two groups with (16) participants in each group. Group A will be given Klapp method exercises to the participant for a period of 1 month twice in a week for 50min. Group B will be given printed information on an at-home exercise program, such, posture correction, corrective exercises and breathing exercises. They will be asked to perform the exercises twice weekly during the study and follow-up period. All these sessions will be of 50 minute for 2 session per week for 4 weeks. Pre and post assessment of pain, pain will be assessed by visual analogue scale, posture will be evaluated by inclinometer, self-efficacy breast feeding will be assessed self-efficacy breastfeeding scale (BSES-SF). Data will be analyzed by using SPSS version 26.0

ELIGIBILITY:
Inclusion Criteria:

* Primiparous females
* Female who had C-Section
* Lactating females (females who have had feed their babies for last 6 months)
* Pain in neck (pain score 4-6 in visual analogue scale)
* Female with kyphotic angle greater than 45 degrees (assess by inclinometer)

Exclusion Criteria:

* history of orthopedic surgery (spinal fusion)
* orthopedic disorder (disk degeneration, osteoporosis)
* history of vertebral fracture
* Female who had given vaginal birth
* Breast feeding issues (lactation failure, nipple failure)

Ages: 22 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — breast feeding females with kyphotic posture
Enrollment: 32 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4th week
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. moderate to good reliability for disability in patients with chronic musculoskeletal pain VAS is widely used as a measure of pain intensity in globally. It has been shown that VAS is valid, reliable and interval scale. The majority of the studies showed that visual analogue scale is a valid and reliable scale. . High reliability when it is used for acute musculoskeletal pain and ICC = 0.99 [95%CI 0.989 to 0.992], and moderate to good reliability for disability in patients with chronic musculoskeletal pain. Also, it is an interval scale. So, in clinical practice we can use this scale in case of measurement as an outcome measure tool.
inclinometer | 4th week
  The gravity-dependent (analogue) inclinometer produces angles that are comparable to the modified Cobb angle obtained from radiographs, establishing its criterion validity as a safe clinical tool for measuring thoracic kyphosis. Inclinometer has high validity with (r=0.85-0.95) and high inter-rater reliability (ICC=0.85-0.98)
Self-efficacy breast feeding scale (BSES-S F questionnaire) | 4th week
  Breastfeeding self-efficacy is defined as a mother's confidence in ability to breastfeed and predicts "whether a mother chooses to breastfeed, how much effort she will expend, whether she will persevere in her attempts until mastery is achieved, whether she will have self enhancing or self-defeating thought patterns, and how she will emotionally respond to breastfeeding difficulties" BSES (n = 5 studies) or BSES-SF (n = 36studies) among demographically or culturally diverse populations. All versions of the instrument demonstrated good reliability, with Cronbach's alphas ranging from .72 to .97

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Civil hospital and Al-siddique hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zappala M, Lightbourne S, Heneghan NR. The relationship between thoracic kyphosis and age, and normative values across age groups: a systematic review of healthy adults. J Orthop Surg Res. 2021 Jul 9;16(1):447. doi: 10.1186/s13018-021-02592-2. PMID 34243795
- [Background] Zanguie H, Yousefi M, Ilbiegi S, Pezeshk AF. Validity and Reliability of Non Invasive Methods for Evaluating Kyphosis and Lordosis Curvatures: A Literature Review. Journal of Modern Rehabilitation. 2023
- [Background] Shafshak TS, Elnemr R. The Visual Analogue Scale Versus Numerical Rating Scale in Measuring Pain Severity and Predicting Disability in Low Back Pain. J Clin Rheumatol. 2021 Oct 1;27(7):282-285. doi: 10.1097/RHU.0000000000001320. PMID 31985722
- [Background] Sebaaly A, Silvestre C, Rizkallah M, Grobost P, Chevillotte T, Kharrat K, Roussouly P. Revisiting thoracic kyphosis: a normative description of the thoracic sagittal curve in an asymptomatic population. Eur Spine J. 2021 May;30(5):1184-1189. doi: 10.1007/s00586-020-06670-7. Epub 2020 Nov 22. PMID 33222002
- [Background] Urrutia J, Besa P, Narvaez F, Meissner-Haecker A, Rios C, Piza C. Mid and lower thoracic kyphosis changes during adulthood: the influence of age, sex and thoracic coronal curvature. Arch Orthop Trauma Surg. 2022 Aug;142(8):1731-1737. doi: 10.1007/s00402-021-03798-z. Epub 2021 Feb 5. PMID 33544182